CLINICAL TRIAL: NCT01544699
Title: Impact of Non-invasive Brain Stimulation on Motor Recuperation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Pr Yves Vandermeeren, MD, PhD, Professor, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B039201212957(2)
Record Dates: First submitted 2012-02-10; First posted 2012-03-06 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Stroke
Keywords: stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: no change
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: no change
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real stimulation (Active Comparator): real tDCS (well, that's the way it is I am not gonna change it)
  Interventions: Device: tDCS (ELDITH)
- Sham (Sham Comparator): sham tDCS
  Interventions: Device: tDCS (ELDITH)

INTERVENTIONS:
Device: tDCS (ELDITH) — tdcs (ELDITH, Neuroconn, Ilmenau, Germany) transcranial direct current stimulation

SUMMARY:
tDCS (transcranial direct current stimulation) will be used in chronic stroke patients to improve a variety of functions with superior or inferior limb.

DETAILED DESCRIPTION:
tDCS will be used in chronic stroke patients to improve a variety of functions such as motor functions with superior or inferior limb.

tDCS will be applied in a placebo-controlled, double-blind, randomised fashion. Behavioural data will be collected before and after tDCS, as well as brain functional imaging data.

ELIGIBILITY:
Inclusion Criteria:

* stroke with at least slight deficit in superior or inferior limb

Exclusion Criteria:

* epilepsy
* contraindication to tDCS and/or to fMRI
* presence of metal in the head
* inability to understand/complete behavioural tasks
* chronic intake of alcohol or recreative drugs
* major health condition
* presence of pacemaker
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
change in motor function before/after tDCS | Baseline (>6 months after stroke), immediately after intervention (30min of tDCS), 10-20-30-40-50-60 min after intervention; long-term after intervention : 1-2-3-4 weeks
  Motor performance improvement with inferior or superior limb

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, CHU Mont-Godinne, Yvoir, Namur,, Belgium

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411